CLINICAL TRIAL: NCT04779229
Title: Linking a Pediatric Healthcare Advance With a Task-Shifting Approach to Optimize Juvenile Justice Outcomes
Brief Title: Leveraging Evidence to Activate Parents
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Responsible Party: Principal Investigator, Mike McCart, Senior Research Scientist, Oregon Social Learning Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DA050669 (NIH)
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Substance Use
Keywords: Substance Use; Delinquency; Parents; Adolescents
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Activation (Experimental): This group of JPOs will deliver Parent Activation as a service to the juveniles and families on their caseloads.
  Interventions: Behavioral: Parent Activation
- Usual Services (Active Comparator): This group of JPOs will deliver services as usual to the juveniles and families on their caseloads.
  Interventions: Behavioral: Usual Services

INTERVENTIONS:
Behavioral: Parent Activation — Parent Activation (PA) is comprised of concrete social learning theory steps (i.e., direct instruction, modeling, practice opportunities, and reinforcement) that aim to enhance a parent's confidence, knowledge, and ability to manage his/her child's health. PA is applicable across a range of conditions, including behavioral and psychiatric problems, and it can be delivered by varied providers, including paraprofessionals.
  Arms: Parent Activation
Behavioral: Usual Services — This intervention refers to the typical techniques that JPOs employ to monitor the juveniles on their caseloads (e.g., regular meetings with youth and parents to ensure the youth is following conditions of probation and issuing swift sanctions [community service; detention] if conditions are not being followed).
  Arms: Usual Services

SUMMARY:
The juvenile justice (JJ) system serves over a million cases every year and represents the primary referral source for treatment of substance use and antisocial behavior in youth. However, engagement of the JJ population in treatment is alarmingly low; further, rural communities have neither access to evidence-based practices (EBPs) nor the finances and treatment infrastructure to support their delivery. However, using an innovation called task-shifting, juvenile probation/parole officers in rural communities might be able to deliver a central change mechanism for EBPs (parent activation), with the ultimate goal of improving JJ youth outcomes.

DETAILED DESCRIPTION:
Juvenile justice (JJ) is the public service system most impacted by alcohol and other drug (AOD) use in youth, and outcomes for these youth, their families, and society are grave. Thus, delivery of effective interventions with JJ youth is of considerable importance. The evidence-based practices (EBPs) with the strongest outcomes for JJ youth are family-based, but many communities do not have the resources to support their delivery. This is particularly true in rural areas where AOD treatment resources are scarce. Further, even when communities can support a family-based EBP, JJ youth face barriers to treatment participation. Indeed, JJ youth are routinely referred for treatment, but data indicate less than 1 in 5 actually receive treatment. Juvenile probation/parole officers (JPOs) are on the front line of this crisis. This workforce is in every community across the nation and routinely interfaces with JJ youth to try to achieve positive outcomes. However, JPOs often face limited options for treatment referrals; further, they do not have the time or training to deliver one of the full-scale, family-based EBPs. As a consequence, JPOs try to manage the behavior of their probationers with a small menu of youth-based interventions that have limited success (e.g., structured sanctions). One strategy for achieving better outcomes in low-resourced, rural settings that cannot deploy a full-scale EBP, called task-shifting, involves redistribution of tasks downstream to an indigenous workforce that has less training. Importantly, reviews indicate that the leading EBPs for JJ youth share a common change mechanism: activation of parents. Thus, while the family-based EBPs cannot be task-shifted, perhaps the central change mechanism of these EBPs (parent activation) can be shifted downstream to enhance JPO practice. JJ leaders already cite improved parent engagement as a top priority, but it is also one of the most challenging problems facing the JJ system. Fortuitously, within pediatric healthcare services, there is an effective intervention called parent activation (PA) comprised of concrete tasks by healthcare service providers to better engage and motivate parents of at-risk youth. PA has been delivered by clinicians and also by paraprofessionals. Thus, this healthcare service advance might be primed for use by JPOs to activate parents and achieve more positive JJ youth outcomes. The proposed stepped-wedge cluster randomized trial investigates the use and impact of PA by JPOs across 32+ rural counties. Aims are to: (1) determine the capacity of JPOs to deliver PA within JJ services, (2) examine impact of PA delivery on de-identified family outcomes, and (3) examine implementation outcomes, assessed via the Stages of Implementation Completion, for PA in the JJ service system, including JPO inner context variables that might impact implementation. In a context where the nation's behavioral healthcare service system is struggling to meet the needs of JJ youth, JPOs across the nation, and particularly in rural communities, are positioned to make a large impact via use of an advance from pediatric healthcare services.

ELIGIBILITY:
Inclusion Criteria:

* Any juvenile probation/parole officer working in a participating county in Idaho or Oregon who consents to participate.

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline scores compared to 36 months post-Baseline on fidelity to Parent Activation (measured at Baseline, End of Usual Services phase, every 3 months for 9 months, and then every 6 months until 36 months post-Baseline). | Baseline to 36 months
  Fidelity to Parent Activation techniques by JPOs as measured using Standardized Patient Assessments (Observational coding of video recordings with trained actors).
Changes in number and severity of criminal charges in de-identified youth records from Baseline compared with 36 months post-Baseline. | Baseline to 36 months
  The number and severity of criminal charges measured by de-identified archival arrest records obtained from Idaho and Oregon state justice databases.

SECONDARY OUTCOMES:
Changes from Baseline in attitudes towards Evidence-Based practices compared to 36 months post-Baseline (measured at 0, 6, 12, 18, 24, 30, and 36 months). | Baseline to 36 months
  Ratings on attitudes towards evidence-based practices as measured by the Evidence-Based Practice Attitude Scale (Self-report completed by the JPOs).
Changes from Baseline in perceived burnout compared to 36 months post-Baseline (measured at 0, 6, 12, 18, 24, 30, and 36 months). | Baseline to 36 months
  Ratings on perceived levels of burnout as measured by the Maslach Burnout Inventory - Human Services Survey (Self-report completed by the JPOs).
Changes from Baseline in perceived agency support of evidence-based practices implementation compared to 36 months post-Baseline (measured at 0, 6, 12, 18, 24, 30, and 36 months). | Baseline to 36 months
  Ratings on perceived agency/county level of support for the implementation of evidence-based practices as measured by the Implementation Climate Survey (Self-report completed by the JPOs).
Changes from Baseline in perceived processes and outcomes between JPOs and the researchers compared to 36 months post-Baseline (measured at 0, 6, 12, 18, 24, 30, and 36 months). | Baseline to 36 months
  Ratings on perceived processes and outputs between the JPOs and the researchers as measured by the Cultural Exchange Inventory (Self-report completed by the JPOs).
Changes from Baseline in de-identified family outcomes (parent attendance and the number of positive youth drug screens) compared to 36 months post-Baseline (measured biweekly for 36 months). | Baseline to 36 months
  De-identified family outcomes (parent attendance and youth drug screen results) at JPO appointments as measured by the Intensive Longitudinal Data Collection Survey created by the researchers (Self-report completed by the JPOs and separately, de-identified parents).
Stage of Implementation reached by 36 months post-Baseline (measured biweekly for 36 months). | Baseline to 36 months
  Dates of implementation milestones of Parent Activation in a county as measured by the Stages of Implementation Completion (Observational codes completed by the researchers).
Changes from Baseline in perceived parent self-efficacy compared to 36 months post-Baseline (measured biweekly for 36 months). | Baseline to 36 months
  Ratings on perceived self-efficacy in parenting measured by the Parent Self-Agency Measure (Self-report completed by de-identified parents attending juvenile probation appointments).

CONTACTS AND LOCATIONS:
Overall Officials: Michael McCart, Ph.D., Principal Investigator — Oregon Social Learning Center
Locations (1):
- Oregon Social Learning Center, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No